CLINICAL TRIAL: NCT01122407
Title: Obesity, Hypertension in African American Women, Neuro-metabolic Mechanism
Brief Title: Pathophysiology of Cardiometabolic Risk Factors in African Americans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Cyndya Shibao, Assistant Professor of Medicine, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 091282; K23HL103976-06 (NIH)
Record Dates: First submitted 2010-05-10; First posted 2010-05-13 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Obesity; Hypertension
MeSH Terms: conditions — Obesity; Hypertension | interventions — omega-N-Methylarginine; Trimethaphan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- trimethaphan (Experimental): Trimethaphan infusion doses of 4 mg/min
  Interventions: Drug: Trimethaphan
- Trimethaphan plus L-NMMA (Experimental): Trimethaphan infusion 4 mg/min L-NMMA (L-NG-monomethyl Arginine citrate) infusion 250 mpg/kg/min A small group of arm 1 will receive both drugs.
  Interventions: Drug: L-NMMA; Drug: Trimethaphan

INTERVENTIONS:
Drug: L-NMMA — L-NMMA 250 ug/Kg/min
  Arms: Trimethaphan plus L-NMMA
Drug: Trimethaphan — Will infuse trimethaphan for until complete autonomic blockade is achieved.

SUMMARY:
The overall goal of this proposal is to determine the autonomic and nitric oxide contribution in the pathogenesis of hypertension and insulin resistance in obese African American women. For this purpose we will use two non-FDA approved drugs:

Trimethaphan IND# 63826 Approval date 12/20/2001 L-NMMA IND# 41735 Approval date 09/1993

DETAILED DESCRIPTION:
The overall goal of this proposal is to determine the autonomic and nitric oxide contribution in the pathogenesis of hypertension and insulin resistance in obese African American women.

Each year cardiovascular disease causes the deaths of approximately 54,000 African American women in the United States.Obesity, hypertension and insulin resistance are more prevalent among African American women as compared to men and Caucasians. These conditions put them at increased risk for the development of diabetes mellitus and cardiovascular disease.

Obesity is associated with increased sympathetic nervous system activity. A positive linear association has been consistently reported between body fat and muscle sympathetic nerve activity (MSNA), a direct measurement of baroreflex modulated vasoconstrictive sympathetic outflow. We and others have reported that in Caucasians this increased sympathetic activation contributes to obesity-associated hypertension. Our preliminary data in African American women indicates that for the same body mass index (BMI), African American women have lower autonomic contribution to blood pressure than Caucasians. We also found important differences in body composition with African American women having less fat mass. When total fat mass is analyzed based on its different components, visceral fat has shown to be a more metabolic active tissue than subcutaneous fat mass, and correlates with sympathetic activity better than any other indices of obesity. Therefore, in specific aim 1a, we propose to test the hypothesis that visceral fat mass modulates the contribution of the autonomic nervous system to blood pressure in obese African American women.

If the autonomic nervous system does not contribute to obesity-associated hypertension in African American women, then what causes these racial differences?. Other pathways involved in blood pressure regulation, such as nitric oxide, might be altered in this group. Several studies have reported that, compared to Caucasians, African Americans have decreased nitric oxide function in isolated vascular beds. The significance of these findings on blood pressure regulation is unknown. We have implemented in our laboratory, new approaches to isolate the contribution of nitric oxide (NO) to blood pressure, by blocking autonomic ganglia neurotransmission with trimethaphan and the production of NO with a nitric oxide synthase inhibitor. This paradigm allows us to define nitric oxide function in the absence of baroreflex buffering or interactions with the autonomic nervous system. In specific aim 1b, we propose to test the hypothesis that obese African American women have impaired NO contribution to blood pressure as part of the pathogenesis of hypertension in this group.

ELIGIBILITY:
Inclusion Criteria:

Race will be self-defined, but only subjects who report both parents of the same race will be included.

All subjects will be pre-menopausal. Age 30-50 years old. We will recruit subjects with wide range of BMI 30-45 kg/m2. Both hypertensives and non-hypertensives will be recruited Hypertension will be defined as a seated blood pressure >130/85 determined in at least two occasions, and therefore, includes patients with "pre-hypertension".

Subjects will be required to have a negative serum/urine pregnancy test. In addition, they will be asked to use a reliable contraceptive method prior to enrollment as determined by the PI (Dr. Cyndya Shibao)

Exclusion Criteria:

Previous allergic reactions to any of the study medications (trimethaphan, L-NMMA, phenylephrine) or inability to take study medications as prescribed during the course of the study.

Use of pacemaker or any metal implant NOT COMPATIBLE WITH MRI (artificial heart valves, implanted drug infusion ports, artificial limb, implanted nerve stimulator, metal pins, screws, plates, surgical staples).

Type 1 or 2 diabetes mellitus as defined by a fasting glucose of 126 mg/dl or greater or the use of anti-diabetic medication.

Cardiovascular disease such as myocardial infarction within 6 months prior to enrollment, presence of angina pectoris, significant arrhythmia, congestive heart failure (LV hypertrophy acceptable), deep vein thrombosis, pulmonary embolism, second or third degree heart block, mitral valve stenosis, aortic stenosis or hypertrophic cardiomyopathy.

History of smoking or current smokers. Significant weight change >5% from baseline in the past three months. Pregnancy or breast-feeding. History of serious neurological disease such as cerebral hemorrhage stroke, transient ischemic attack.

History or presence of immunological or hematological disorders. Clinical significant gastrointestinal impairment that could interfere with drug absorption.

Impaired hepatic function (aspartate amino transaminase [AST] and/or alanine amino transaminase [ALT] >1.5X upper limit of normal range).

Impaired renal function (estimated glomerular filtration rate (eGFR) of <60mL/min).

Any underlying or acute disease requiring regular medication which could possibly pose a threat to the subject or make implementation of the protocol or interpretation of the study results difficult.

History of alcohol or drug abuse. Mental conditions rendering the subject unable to understand the nature, scope and possible consequences of the study.

Inability to comply with the protocol, e.g. uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study.

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2010-01; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
change in systolic blood pressure in response to trimethaphan, as a measurement of the tonic sympathetic contribution to blood pressure. | 30 minutes after initiation of Trimethaphan infusion
  Will infuse trimethaphan for until complete autonomic blockade is achieved.

SECONDARY OUTCOMES:
increase in systolic blood pressure induced by NOS inhibition with 250 ug/kg/min L-NMMA during autonomic withdrawal with trimethaphan. | within 30 minutes
  After achieving complete autonomic blockade will infuse L-NMMA.

CONTACTS AND LOCATIONS:
Overall Officials: Cyndya Shibao, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rahman S, Gamboa A, Saleem M, Kulapatana S, Diedrich A, Biaggioni I, Kirabo A, Shibao CA. Complete autonomic blockade reveals nitric oxide contribution to blood pressure regulation in obese Black women. Clin Auton Res. 2024 Aug;34(4):427-436. doi: 10.1007/s10286-024-01050-3. Epub 2024 Aug 1. PMID 39090323